CLINICAL TRIAL: NCT05355233
Title: Comparative Effects of Bebo Concept and Diaphragmatic Breathing Technique on Stress Incontinence in Females After Vaginal Birth
Brief Title: Comparative Effects of Bebo Concept and Diaphragmatic Breathing Technique on Stress Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/21/0524
Record Dates: First submitted 2022-04-15; First posted 2022-05-02 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Urinary Incontinence
Keywords: Bebo Concept, diaphragmatic breathing, vaginal delivery
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bebo concept (Experimental): it is a technique to deal urinary incontinence
  Interventions: Other: bebo concept
- diaphragmatic breathing (Experimental): breathing technique to strengthen core muscles
  Interventions: Other: diaphragmatic breathing

INTERVENTIONS:
Other: bebo concept — techniques to remove urinary incontinence
  Arms: bebo concept
Other: diaphragmatic breathing — techniques to remove urinary incontinence
  Arms: diaphragmatic breathing

SUMMARY:
Pelvic floor muscle dysfunctions can lead to urinary incontinence, a condition which often affects female both during pregnancy and after childbirth. As a result of this, certain exercises are recommended during and after pregnancy to prevent and treat this incontinence, and the BeBo Concept is one of these methods used to prevent pelvic floor muscle dysfunction. Urinary incontinence among female is considered a social disease, which may affect up to 20-60% of the population of female over 18 years of age. The strength and endurance of the pelvic floor muscles decrease significantly after the first delivery. Research shows that 65% of female with urinary incontinence remember that the first episode of urine loss occurred during pregnancy or in the puerperium. Prior to the study, all participants will be informed of the purpose and method of Conducting the research. . A 6-week physical therapy program according to the BeBo Pelvic Floor Training Concept. Individual meetings will be twice a week, each lasting 60 min. Each meeting will consist of a theoretical part lasting up to 10 min and a practical part lasting about 50 min. In addition, each participant will receive a set of exercises to be performed at home once daily. For the experimental group, In the first week (meetings 1 and 2), the homework will include the following activities: concentration on the pelvic floor muscles and becoming aware of them in various body positions, mobilization of the pelvis in a sitting position on a chair- 10x, lying on the back with bent legs and activation of PFM with exhalation, inhalation- relaxation-10x, balance exercise, standing on one leg, 10 s each leg, and so on to 6 weeks. Treatment protocol for Control Group (Diaphragmatic Breathing), Exercise programs will consist of 1 set of contractions per day and each set will include 30 repetitions for 6 weeks. Female will be asked to complete forms before starting the program and again at the end of the 6-week program.

DETAILED DESCRIPTION:
Pelvic floor muscle dysfunctions can lead to urinary incontinence, a condition which often affects female both during pregnancy and after childbirth. As a result of this, certain exercises are recommended during and after pregnancy to prevent and treat this incontinence, and the BeBo Concept is one of these methods used to prevent pelvic floor muscle dysfunction. Urinary incontinence among female is considered a social disease, which may affect up to 20-60% of the population of female over 18 years of age. The strength and endurance of the pelvic floor muscles decrease significantly after the first delivery. Research shows that 65% of female with urinary incontinence remember that the first episode of urine loss occurred during pregnancy or in the puerperium. Prior to the study, all participants will be informed of the purpose and method of Conducting the research. Each of them will sign an informed consent release to participate in the project and to process personal data for scientific purposes. We confirm that all research will be performed in accordance with relevant guidelines and regulations. A 6-week physical therapy program according to the BeBo Pelvic Floor Training Concept. Individual meetings will be twice a week, each lasting 60 min. Each meeting will consist of a theoretical part lasting up to 10 min and a practical part lasting about 50 min. In addition, each participant will receive a set of exercises to be performed at home once daily. For the experimental group, In the first week (meetings 1 and 2), the homework will include the following activities: concentration on the pelvic floor muscles and becoming aware of them in various body positions, mobilization of the pelvis in a sitting position on a chair- 10x, lying on the back with bent legs and activation of PFM with exhalation, inhalation- relaxation-10x, balance exercise, standing on one leg, 10 s each leg, and so on to 6 weeks. Treatment protocol for Control Group (Diaphragmatic Breathing), Exercise programs will consist of 1 set of contractions per day and each set will include 30 repetitions for 6 weeks. Female will be asked to complete forms before starting the program and again at the end of the 6-week program.

ELIGIBILITY:
Inclusion Criteria:

* • Primiparous females with a single pregnancy

  * 20-40 years old
  * Delivery between 37 and 42 weeks of pregnancy
  * 6 to 8 weeks after natural childbirth
  * No contraindications to exercise stated by an obstetrician

Exclusion Criteria:

* Multiple pregnancy

  * Caesarean delivery
  * Postpartum complications in the form of: separation of the pubic symphysis and sacroiliac joints thrombophlebitis, 3rd and 4th degree of perineal rupture, urinary tract or vaginal infections/infections during the experiment, 3rd and 4th degree of pelvic organ prolapse, 3rd degree of stress urinary incontinence or overactive bladder diagnosed before pregnancy, gynecological surgeries, spine operations, pelvic and spine fractures, injuries, operations on the lower limbs 12 months or less previous to the study, diseases of the nervous system, e.g. MS, stroke, respiratory diseases, diabetes, cancer, rheumatic diseases.
  * Refusal to participate in the study

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 66 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
UDI-6 (Urinary distress inventory, short form) | 6 months
  Urogenital Distress Inventory-6 (UDI-6) used to diagnose individuals with urinary incontinence
ICIQ-SF Questionnaire The ICIQ-UI Short Form | 6 months
  The ICIQ-UI Short Form is a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women in research and clinical practice across the world. This short and simple questionnaire is also of use to general practitioners and clinicians in both primary and secondary care institutions to screen for incontinence, to obtain a brief yet comprehensive summary of the level, impact and perceived cause of symptoms of incontinence and to facilitate patient-clinician discussions.
Palpation perfect test | 6 months
  It is performed by inserting a finger (or fingers) into the vaginal cavity. Pelvic floor muscle contraction can be felt and the therapist is looking for both a squeeze and lift.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rabiya Noor, PhD, Study Chair — Riphah International University
Locations (1):
- Jinah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toprak N, Sen S, Varhan B. The role of diaphragmatic breathing exercise on urinary incontinence treatment: A pilot study. J Bodyw Mov Ther. 2022 Jan;29:146-153. doi: 10.1016/j.jbmt.2021.10.002. Epub 2021 Oct 20. PMID 35248263
- [Background] Sniezek A, Czechowska D, Curylo M, Glodzik J, Szymanowski P, Rojek A, Marchewka A. Physiotherapy according to the BeBo Concept as prophylaxis and treatment of urinary incontinence in women after natural childbirth. Sci Rep. 2021 Sep 10;11(1):18096. doi: 10.1038/s41598-021-96550-x. PMID 34508116